CLINICAL TRIAL: NCT01306162
Title: Relative Bioavailability of a Single Dose of 150 mg Dabigatran Etexilate (Capsule) When Administered Alone or in Combination With a Single Dose of 400 mg Dronedarone Tablet) or in Combination With 400 mg Bid Dronedarone (Tablet) at Steady State in Healthy Male and Female Volunteers (an Open Label, Randomised, Four-sequence, Two Period Cross-over, Phase I Study)
Brief Title: Drug Interaction Study With Dabigatran Etexilate and Dronedarone in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.112; 2010-024009-11 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Dronedarone

ARMS (5):
- A: Dabigatran alone (Reference) (Experimental): Capsule, oral administration with 240 mL water
  Interventions: Drug: Dabigatran etexilate
- B: Dabigatran plus Dronedarone (Test) (Experimental): Capsule and Tablets, oral administration with 240 mL water
  Interventions: Drug: Dabigatran etexilate plus dronedarone
- C: Dabigatran plus Dronedarone (Test) (Experimental): Capsule and Tablets, oral administration with 240 mL water
  Interventions: Drug: Dabigatran etexilate plus dronedarone
- D: Dabigatran plus Dronedarone (Test) (Experimental): Capsule and Tablets, oral administration with 240 mL water
  Interventions: Drug: Dabigatran etexilate plus dronedarone
- E: Dabigatran plus Dronedarone (Test) (Experimental): Capsule and Tablets, oral administration with 240 mL water
  Interventions: Drug: Dabigatran etexilate plus dronedarone

INTERVENTIONS:
Drug: Dabigatran etexilate plus dronedarone — dabigatran etexilate 150 mg plus dronedarone 400 mg as single dose
  Arms: B: Dabigatran plus Dronedarone (Test)
Drug: Dabigatran etexilate — 150 mg as single dose
  Arms: A: Dabigatran alone (Reference)
Drug: Dabigatran etexilate plus dronedarone — dabigatran etexilate 150 mg plus dronedarone 400 mg as single dose (staggered administration)
  Arms: C: Dabigatran plus Dronedarone (Test)
Drug: Dabigatran etexilate plus dronedarone — dabigatran etexilate 150 mg single dose plus dronedarone 400 mg bid
  Arms: D: Dabigatran plus Dronedarone (Test)
Drug: Dabigatran etexilate plus dronedarone — dabigatran etexilate 150 mg single dose plus dronedarone 400 mg bid (staggered administration)
  Arms: E: Dabigatran plus Dronedarone (Test)

SUMMARY:
The objective of the study is to assess the relative bioavailability of a single dose of dabigatran after concomitant multiple oral administration of dronedarone with the aim to investigate whether and to what extent the P-gp inhibitor dronedarone affects pharmacokinetic parameters of dabigatran when administered to healthy subjects

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.112.1 Boehringer Ingelheim Investigational Site, Ulm, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this crossover study, subjects were randomly assigned to one of the 4 sequences, but with 5 treatments. In general terms ABDE,ACED,BDEA,CEDA. There were four subjects in Trt E who took Dronedarone mistakenly in place of Dabigatran. These are presented separately for adverse events.
Groups:
- TrtA -- TrtB -- TrtD -- TrtE: Dabigatran 150mg (Trt. A), followed by Dabigatran 150mg + Dronedarone 400mg given simultaneously (Trt. B), followed by Dabigatran 150mg + Dronedarone 400mg bid given simultaneously (Trt. D), followed by Dabigatran 150mg + Dronedarone 400mg bid given 2h later (Trt. E)
- TrtA -- TrtC -- TrtE -- TrtD: Dabigatran 150mg (Trt. A), followed by Dabigatran 150mg + Dronedarone 400mg given 2h later (Trt. C), followed by Dabigatran 150mg + Dronedarone 400mg bid given 2h later (Trt. E), followed by Dabigatran 150mg + Dronedarone 400mg bid given simultaneously (Trt. D)
- TrtB -- TrtD -- TrtE -- TrtA: Dabigatran 150mg + Dronedarone 400mg given simultaneously (Trt. B), followed by Dabigatran 150mg + Dronedarone 400mg bid given simultaneously (Trt. D), followed by Dabigatran 150mg + Dronedarone 400mg bid given 2h later (Trt. E), followed by Dabigatran 150mg (Trt. A)
- TrtC -- TrtE -- TrtD -- TrtA: Dabigatran 150mg + Dronedarone 400mg given 2h later (Trt. C), followed by Dabigatran 150mg + Dronedarone 400mg bid given 2h later (Trt. E), followed by Dabigatran 150mg + Dronedarone 400mg bid given simultaneously (Trt. D), followed by Dabigatran 150mg (Trt. A)
Period: Period 1
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Washout 1
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA
Started | 9 (Treatment A was followed by a washout period of at least 96 hours.) | 9 (Treatment A was followed by a washout period of at least 96 hours.) | 9 (No washout period. Treatment D followed directly after treatment B.) | 8 (No washout period.Treatment E followed directly after treatment C.)
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 1 | 0 | 0
Not completed — Non-compliance to protocol | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA
Started | 9 (No washout phase after Period 2.) | 8 (No washout phase after Period 2.) | 9 (No washout phase after Period 2.) | 8 (No washout phase after Period 2.)
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA
Started | 9 | 8 | 9 | 8
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout 2
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA
Started | 9 (No washout period. Treatment E followed directly after treatment D.) | 8 (No washout period. Treatment D followed directly after treatment E.) | 9 (The last dose of Dronedarone was followed by a washout period of at least 10 days.) | 8 (The last dose of Dronedarone was followed by a washout period of at least 10 days.)
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA
Started | 9 | 8 | 9 | 8
Completed | 9 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set contains of all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TrtA -- TrtB -- TrtD -- TrtE | TrtA -- TrtC -- TrtE -- TrtD | TrtB -- TrtD -- TrtE -- TrtA | TrtC -- TrtE -- TrtD -- TrtA | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (10.7) | 37.8 (10.4) | 38.1 (9.7) | 33.3 (7.9) | 35.4 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 2 | 5 | 19
  Male | 2 | 4 | 7 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Total Dabigatran: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of total dabigatran in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: 1 h before drug administration and 0:30, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00, 36:00, 48:00 h after drug administration
Population: Pharmacokinetic (PK) set defined as all subjects randomised, treated and who provided evaluable data for at least one observation for at least one primary endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 150mg DE (TrtA): Dabigatran 150mg
- 150mg DE + 400mg DR (TrtB): Dabigatran 150mg + Dronedarone 400mg given simultaneously
- 150mg DE + 400mg DR 2h Later (TrtC): Dabigatran 150mg + Dronedarone 400mg given 2h later
- 150mg DE + 400mg DR Bid Same Time (TrtD): Dabigatran 150mg + Dronedarone 400mg bid given simultaneously
- 150mg DE + 400mg DR Bid 2h Later (TrtE): Dabigatran 150mg + Dronedarone 400mg bid given 2h later
Arm/Group | 150mg DE (TrtA) | 150mg DE + 400mg DR (TrtB) | 150mg DE + 400mg DR 2h Later (TrtC) | 150mg DE + 400mg DR Bid Same Time (TrtD) | 150mg DE + 400mg DR Bid 2h Later (TrtE)
Number analyzed (Participants) | 35 | 18 | 17 | 34 | 30
ng*hr/mL | 1160 (40.3) | 2520 (27.1) | 1440 (40.3) | 2570 (28.1) | 1510 (32.9)
Statistical Analysis 1: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR (TrtB); 150mg DE + 400mg DR same time (TrtB) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 1.0000, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtB: TrtA (%) = 214, 90% CI 2-sided [191 to 240], Standard Deviation 19.9 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 2: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR 2h Later (TrtC); 150mg DE + 400mg DR 2h later (TrtC) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.6697, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtC: TrtA (%) = 130, 90% CI 2-sided [112 to 151], Standard Deviation 25.0 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 3: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid Same Time (TrtD); 150mg DE + 400mg DR bid same time (TrtD) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9992, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtD: TrtA (%) = 236, 90% CI [173 to 321], Standard Deviation 21.8 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 4: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid 2h Later (TrtE); 150mg DE + 400mg DR bid 2h later (TrtE) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9171, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtE: TrtA (%) = 162, 90% CI 2-sided [119 to 221], Standard Deviation 20.1 — The standard deviation is actually the Geometric coefficient of variation

2. Primary Outcome: Total Dabigatran: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of total dabigatran in plasma, per period.
Time Frame: as for outcome 1
Population: PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 150mg DE (TrtA) | 150mg DE + 400mg DR (TrtB) | 150mg DE + 400mg DR 2h Later (TrtC) | 150mg DE + 400mg DR Bid Same Time (TrtD) | 150mg DE + 400mg DR Bid 2h Later (TrtE)
Number analyzed (Participants) | 35 | 18 | 17 | 34 | 30
ng/mL | 149 (46.0) | 282 (30.1) | 166 (37.5) | 288 (29.9) | 163 (30.9)
Statistical Analysis 1: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR (TrtB); 150mg DE + 400mg DR (TrtB) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9999, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtB: TrtA (%) = 187, 90% CI 2-sided [162 to 215], Standard Deviation 24.3 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 2: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR 2h Later (TrtC); 150mg DE + 400mg DR 2h later (TrtC) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.2207, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtC: TrtA (%) = 115, 90% CI 2-sided [95 to 138], Standard Deviation 31.2 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 3: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid Same Time (TrtD); 150mg DE + 400mg DR bid same time (TrtD) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9946, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtD: TrtA (%) = 225, 90% CI [156 to 326], Standard Deviation 26.1 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 4: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid 2h Later (TrtE); 150mg DE + 400mg DR bid 2h later (TrtE) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.6221, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtE: TrtA (%) = 133, 90% CI 2-sided [94 to 190], Standard Deviation 23.0 — The standard deviation is actually the Geometric coefficient of variation

3. Secondary Outcome: Free Dabigatran: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of free dabigatran in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 1
Population: PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 150mg DE (TrtA) | 150mg DE + 400mg DR (TrtB) | 150mg DE + 400mg DR 2h Later (TrtC) | 150mg DE + 400mg DR Bid Same Time (TrtD) | 150mg DE + 400mg DR Bid 2h Later (TrtE)
Number analyzed (Participants) | 35 | 18 | 17 | 34 | 30
ng*hr/mL | 919 (47.5) | 2110 (27.4) | 1110 (47.2) | 2100 (30.5) | 1260 (36.0)
Statistical Analysis 1: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR (TrtB); 150mg DE + 400mg DR (TrtB) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 1.0000, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtB: TrtA (%) = 214, 90% CI 2-sided [190 to 241], Standard Deviation 20.7 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 2: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR 2h Later (TrtC); 150mg DE + 400mg DR 2h later (TrtC) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.7223, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtC: TrtA (%) = 132, 90% CI 2-sided [113 to 155], Standard Deviation 26.3 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 3: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid Same Time (TrtD); 150mg DE + 400mg DR bid same time (TrtD) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9993, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtD: TrtA (%) = 258, 90% CI [182 to 365], Standard Deviation 24.6 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 4: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid 2h Later (TrtE); 150mg DE + 400mg DR bid 2h later (TrtE) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.8875, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtE: TrtA (%) = 159, 90% CI 2-sided [114 to 222], Standard Deviation 21.5 — The standard deviation is actually the Geometric coefficient of variation

4. Secondary Outcome: Free Dabigatran: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of free dabigatran in plasma, per period.
Time Frame: as for outcome 1
Population: PK set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 150mg DE (TrtA) | 150mg DE + 400mg DR (TrtB) | 150mg DE + 400mg DR 2h Later (TrtC) | 150mg DE + 400mg DR Bid Same Time (TrtD) | 150mg DE + 400mg DR Bid 2h Later (TrtE)
Number analyzed (Participants) | 35 | 18 | 17 | 34 | 30
ng/mL | 126 (48.0) | 239 (27.6) | 133 (40.7) | 241 (29.5) | 138 (34.0)
Statistical Analysis 1: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR (TrtB); 150mg DE + 400mg DR (TrtB) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9998, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtB: TrtA (%) = 180, 90% CI 2-sided [156 to 207], Standard Deviation 24.6 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 2: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR 2h Later (TrtC); 150mg DE + 400mg DR 2h later (TrtC) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.1866, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtC: TrtA (%) = 114, 90% CI 2-sided [95 to 136], Standard Deviation 29.4 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 3: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid Same Time (TrtD); 150mg DE + 400mg DR bid same time (TrtD) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.9958, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtD: TrtA (%) = 234, 90% CI [160 to 340], Standard Deviation 26.7 — The standard deviation is actually the Geometric coefficient of variation
Statistical Analysis 4: Comparison: 150mg DE (TrtA) vs 150mg DE + 400mg DR Bid 2h Later (TrtE); 150mg DE + 400mg DR bid 2h later (TrtE) vs 150mg DE (TrtA); Test type: Non-Inferiority or Equivalence — Bioavailability; p = 0.5164, ANOVA — p-value for geometric mean ratio being outside interval 80% to 125%; ANOVA with sequence, period and treatment as fixed effects and subject within sequence as random effect; Geometric mean ratio TrtE: TrtA (%) = 126, 90% CI 2-sided [89 to 179], Standard Deviation 22.6 — The standard deviation is actually the Geometric coefficient of variation

ADVERSE EVENTS:
Time Frame: 14 days
Groups:
- 400mg DR + 400mg DR Bid 2h Later (TrtE2): Dronedarone 400mg + Dronedarone 400mg bid given 2h later
Arm/Group | 150mg DE (TrtA) | 150mg DE + 400mg DR (TrtB) | 150mg DE + 400mg DR 2h Later (TrtC) | 150mg DE + 400mg DR Bid Same Time (TrtD) | 150mg DE + 400mg DR Bid 2h Later (TrtE) | 400mg DR + 400mg DR Bid 2h Later (TrtE2)
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/18 | 0/17 | 0/34 | 0/30 | 0/4
Other Adverse Events (participants affected / at risk) | 3/35 | 6/18 | 5/17 | 5/34 | 3/30 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 150mg DE (TrtA) (N=35) | 150mg DE + 400mg DR (TrtB) (N=18) | 150mg DE + 400mg DR 2h Later (TrtC) (N=17) | 150mg DE + 400mg DR Bid Same Time (TrtD) (N=34) | 150mg DE + 400mg DR Bid 2h Later (TrtE) (N=30) | 400mg DR + 400mg DR Bid 2h Later (TrtE2) (N=4)
Listless (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 4 | 1 | 2 | 2 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.